CLINICAL TRIAL: NCT04393766
Title: Effectiveness of Prophylactic Intrathecal Normal Saline for Prevention of Post Dural Puncture Headache in Women Undergoing Cesarean Section Under Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: Prophylactic Intrathecal Normal Saline for Prevention of Post Dural Puncture Headache in Women Undergoing Cesarean Section Under Spinal Anesthesia
Acronym: PDPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dilla University (Other)
Responsible Party: Principal Investigator, Semagn Mekonnen, Assistant professor of Anesthesiology, Dilla University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0014/19-11
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: PDPH
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: after random generation sequence, the list of 152 were sealed with envelope which later opened by research assistance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal saline (Experimental)
  Interventions: Drug: Normal Saline
- non normal saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Normal Saline — normal saline(crystalloids)

SUMMARY:
The rates of cesarean section are increasing worldwide despite ten to fifteen percent of World Health Organization recommendation and from which 80-90% of cesarean sections are performed with spinal anesthesia. Post Dural Puncture Headache is the commonest complications associated with spinal anesthesia with prevalence as high as forty percent in Ethiopia. Body of evidence revealed that Conservative managements failed to show significant benefit and epidural needle and catheter techniques didn't provide conclusive evidences. On the other hand, intrathecal injection of normal saline is very safe, simple technique and cost effective in resource limited set up but it is not well examined on its efficacy and safety profiles. The main objective of the study is to assess of efficacy and safety of prophylactic Intrathecal Normal Saline for prevention of Post Dural Puncture Headache in women undergoing cesarean section under spinal anesthesia. After Obtaining Ethical clearance from IRB, a Randomized Controlled Trial study will be conducted in Dilla University Referral Hospital from december2019 to December, 2020. 152 mothers scheduled caesarean section under spinal anesthesia fulfilling the inclusion criteria will be allocated into two groups randomly with random sequence generated list obtained from R package (Random Allocation Rule function) software version 3.6.

DETAILED DESCRIPTION:
The rates of cesarean section are increasing worldwide despite ten to fifteen percent of World Health Organization recommendation and from which 80-90% of cesarean sections are performed with spinal anesthesia. Post Dural Puncture Headache is the commonest complications associated with spinal anesthesia with prevalence as high as forty percent in Ethiopia. Body of evidence revealed that Conservative managements failed to show significant benefit and epidural needle and catheter techniques didn't provide conclusive evidences. On the other hand, intrathecal injection of normal saline is very safe, simple technique and cost effective in resource limited set up but it is not well examined on its efficacy and safety profiles. The main objective of the study is to assess of efficacy and safety of prophylactic Intrathecal Normal Saline for prevention of Post Dural Puncture Headache in women undergoing cesarean section under spinal anesthesia.

After Obtaining Ethical clearance from IRB, a Randomized Controlled Trial study will be conducted in Dilla University Referral Hospital from October 2019 to May, 2020. 152 mothers scheduled caesarean section under spinal anesthesia fulfilling the inclusion criteria will be allocated into two groups randomly with random sequence generated list obtained from R package (Random Allocation Rule function) software version 3.6. Data will be entered, cleaned by Epi-info version 7 and imported to Statistical Package for Social Sciences version 22 for analysis. Descriptive statistics will be run to see the overall distribution of the study subjects with regard to the variables under study. Unpaired student's T-test for continuous symmetric data and Mann Whitney U test for non-normally distributed data will be used to see the mean difference between the groups. Categorical data will be analyzed with Chi square and fisher's exact test where appropriate. Survival analysis will be done to estimate the probability having PDPH within five days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists' physical status classification(ASA I and II)
* Term pregnant lady

Exclusion Criteria:

* patient whose ASA status was greater than three
* previous history of PDPH
* previous history of migraine headache
* BMI greater than 25 kg/m2

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of PDPH | for five days postoperatively( 12hrs -5 days)
  occurance of post dural puncture headache
severity of PDPH | 12hrs to 5 days postoperatively
  severity of PDPH will be assessed with validated scale( visual analog score)

SECONDARY OUTCOMES:
peak sensory block | 30 minutes after injection of spinal anesthetics
  sensory block
motor block | 30 minutes after spinal injection
  motor block with bromage score

CONTACTS AND LOCATIONS:
Locations (1):
- Yassin, Addis Ababa, Dilla, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided